CLINICAL TRIAL: NCT07207785
Title: PirtobrUtinib as Frontline Therapy for Elderly Unfit/Frail Patient With MAntle Cell Lymphoma: a Phase II Study of the Fondazione Italiana Linfomi (FIL)
Brief Title: PirtobrUtinib as Frontline Therapy for Elderly Unfit/Frail Patient With MAntle Cell Lymphoma
Acronym: FIL_PUMA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_PUMA
Record Dates: First submitted 2025-09-17; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Mantle Cell Lymphoma
Keywords: mantle cell lymphoma; unfit; frail; monotherapy; pirtobrutinib; Jaypirca
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — pirtobrutinib

STUDY DESIGN:
Intervention Model Description: This is a one-arm phase II study, with a hypothesis of superior efficacy compared to usual/standard clinical approaches.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Pirtobrutinib monotherapy in untreated elderly unfit/frail MCL patients.
  Interventions: Drug: Pirtobrutinib

INTERVENTIONS:
Drug: Pirtobrutinib — Patients will receive pirtrobrutinib at a starting dose of 200 mg once daily (q.d). All treatment will be administered orally and a cycle will be defined as 28 days in length and should be maintained regardless of dose interruptions. Treatment is meant to be administered until tumor progression, unacceptable adverse event, or patient decision for interruption.
  Other Names: Jaypirca

SUMMARY:
This is a prospective, multicenter, phase II study, in elderly patients affected by Mantle cell lymphoma (MCL) defined as unfit/frail according to Simplified Geriatric Assessment (sGA) and previously untreated.

Patients will receive a treatment with Pirtobrutinib monotherapy until tumor progression, unacceptable adverse event, or patient decision for interruption.

DETAILED DESCRIPTION:
After providing written informed consent, patients will be evaluated for eligibility during a 28-day screening period. Patients will receive pirtobrutinib at a starting dose of 200 mg once daily (2 tablets q.d.). All treatment will be administered orally, and a cycle will be defined as 28 days in length and should be maintained regardless of dose interruptions. Treatment is meant to be administered until tumor progression, unacceptable adverse event, or patient decision for interruption.

Responses shall be assessed at month +3, +6 after start of treatment and then every 6 months using the radiologic method of tumor assessment consistent throughout the study and aligned with the baseline method (CT scan or ultrasound echography are acceptable). Positron Emission Tomography (PET) scan is mandatory at baseline and at month +3 after start of treatment to establish tumor response.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented diagnosis of nodal and extranodal mantle cell lymphoma (MCL) as defined in the 2022 edition of the World Health Organization (WHO) classification
2. Availability of biopsy material for central pathology revision and mutational analysis including TP53 (Tumor Protein p53) mutations
3. Age ≥ 70 years
4. Previously untreated MCL
5. Active disease in need of treatment according to clinical practice (patients with leukemic with symptomatic leukemic non nodal disease may be included)
6. Ineligible to standard full-dose induction therapy (i.e. BR, R-CHOP, VR-CAP, RBAC500)
7. sGA assessment performed before starting treatment

   FRAIL patients defined as follows:
   * Age ≥ 80 years
   * Activities of Daily Living (ADL) <6 residual functions and/or
   * Instrumental Activities of Daily Living (IADL) <8 residual functions and/or
   * Cumulative Illness Rating Scale (CIRS): ≥ 1 comorbidity of grade 3-4 or ≥ 5 comorbidities of grade 2

   UNFIT patients defined as follows:
   * Age ≥ 80 years:
   * ADL 6 residual functions and
   * IADL 8 residual functions and
   * CIRS 0 comorbidities of grade 3-4 and <5 comorbidities of grade 2

   or
   * Age < 80 years:
   * ADL < 5 residual functions and/or
   * IADL < 6 residual functions and/or
   * CIRS ≥ 1 comorbidity of grade 3-4 or >8 comorbidities of grade 2
8. Ann Arbor Stage I - IV
9. At least one bi-dimensionally measurable lesion defined as > 1.5 cm in its largest dimension on CT scan
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0- 2
11. Adequate hematologic function (unless caused by bone marrow infiltrate), defined as follows:

    1. Hemoglobin ≥ 8 g/dL (independent of transfusions within 7 days of screening assessment)
    2. White blood cells (WBC) > 2500/mmc with polymorphonuclear (cells) PMN≥750/ mmc) (independent of growth factor support within 7 days of screening assessment)
    3. Platelets count ≥ 50000/mmc (independent of transfusions within 7 days of screening assessment)
12. Adequate renal function:

    * Creatinine clearance ≥ 30 mL/min or
    * Serum creatinine ≤ 2.5 mg /dL
13. Adequate coagulation, defined as activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) and prothrombin (PT) or (international normalized ratio (INR) not greater than 1.5 x upper limit of normal (ULN)
14. Adequate hepatic function:

    * Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) ≤ 3 x the ULN or ≤ 5 x ULN with documented liver involvement
    * Total bilirubin ≤ 1.5 x ULN or ≤ 3 x ULN with documented liver involvement and/or due to Gilbert's Disease
15. Ability and willingness to comply with the study protocol procedure
16. Life expectancy > 6 months
17. The patient is able to take oral medications
18. The patient must give written informed consent
19. Male subjects must use highly effective contraception during sexual contact with a pregnant female or a female of childbearing potential from the start of study treatment and continuing for at least 3 months after the last dose of pirtobrutinib

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible to enroll:

1. Candidate to watch and wait due to indolent presentation
2. Leukemic non-nodal MCL that has stable asymptomatic disease should not be included in this study
3. Histological diagnosis different from MCL or leukemic non-nodal MCL
4. Fit patients according to sGA eligible to standard full dose therapy
5. Candidate or eligible to full-dose Bendamustine+Rituximab (BR), Rituximab + Cyclophosphamide, Hydroxydaunorubicin (doxorubicin), Oncovin (vincristine) e Prednisone (R-CHOP), bortezomib, rituximab, cyclophosphamide, doxorubicin, prednisone (VR-CAP), Rituximab, Bendamustine, Cytarabine (RBAC500) or any other full dose intensive chemotherapy
6. Suspect or clinical evidence of central nervous system (CNS) involvement by lymphoma
7. Contraindication to the use Bruton Tyrosine Kinase Inhibitor (BTKi)
8. HBsAg positivity; HBsAg-negative patients with anti-hepatitis B core antigen (HBc) antibody can be enrolled if Hepatitis B Virus (HBV)-DNA are negative and prophylactic antiviral treatment is provided
9. HIV positivity
10. Active herpes zoster infection; previously infected patients is accepted only with concomitant treatment with Valacyclovir
11. Major surgery within 4 weeks prior to investigation treatment
12. Any history of other malignancies unless in remission and with life expectancy > 2 years prior to study entry except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer
13. Patients who experienced grade ≥ 3 arrhythmia.
14. History of severe bleeding diathesis (major bleeding event) Note: Major bleeding is defined as bleeding having one or more of the following features: potentially life-threatening bleeding with signs or symptoms of hemodynamic compromise; bleeding associated with a decrease in the hemoglobin level of at least 2 g per deciliter; or bleeding in a critical area or organ (e.g., retroperitoneal, intraarticular, pericardial, epidural, or intracranial bleeding or intramuscular bleeding with compartment syndrome)
15. History of stroke or intracranial hemorrhage within 6 months of investigation treatment
16. History of Chimeric Antigen Receptor T-cell therapy (CAR-T) within 60 days of investigation treatment or presence of any of the following, regardless of prior Stem Cell Transplantation (SCT) and/or CAR-T therapy timing:

    1. active graft versus host disease (GVHD);
    2. cytopenia from incomplete blood cell count recovery post-transplant;
    3. need for anti-cytokine therapy for toxicity from CAR-T therapy; residual symptoms of neurotoxicity > Grade 1 from CAR-T therapy;
    4. ongoing immunosuppressive therapy (> 20 mg prednisone or equivalent daily)
17. Evidence of any severe active acute or chronic infection
18. Hepatitis C virus (HCV): positive hepatitis C antibody. If positive hepatitis C antibody result, HCV-RNA is required. Only patients with HCV-RNA negative are accepted.
19. Known active cytomegalovirus (CMV) infection. Unknown or negative status are eligible
20. Clinically significant active malabsorption syndrome or other conditions likely to affect gastrointestinal (GI) absorption of the study drug
21. Evidence of other clinically significant uncontrolled condition(s) including but not limited to, uncontrolled systemic bacterial, viral, fungal or parasitic infection (except for fungal nail infection), or other clinically significant active disease process which in the opinion of the investigator and medical monitor may pose a risk for patient participation. Screening for chronic conditions is not required
22. Active uncontrolled auto-immune cytopenia (e.g., AutoImmune Hemolytic Anemia [AIHA], Idiopathic Thrombocytopenic Purpura [ITP]) for which new therapy was introduced or existing therapy was escalated within the 4 weeks prior to study enrollment to maintain adequate blood counts
23. Significant cardiovascular disease defined as:

    1. unstable angina or acute coronary syndrome within the past 2 months prior to study enrollment
    2. history of myocardial infarction within 3 months prior to study enrollment or
    3. documented left ventricular ejection fraction (LVEF) by any method of ≤ 40% in the 12 months prior to study enrollment
    4. ≥ Grade 3 New York Heart Association (NYHA) functional classification system of heart failure
    5. Uncontrolled or symptomatic arrhythmias
24. Prolongation of the QT interval corrected for heart rate (QTcF) > 470 msec. QTcF is calculated using Fridericia's Formula (QTcF): QTcF = QT/(RR0.33):

    1. Correction of suspected drug-induced QTcF prolongation can be attempted at the investigator's discretion and only if clinically safe to do so with either discontinuation of the offending drug or switch to another drug not known to be associated with QTcF prolongation.
    2. Correction for underlying bundle branch block (BBB) allowed. Note: Patients with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker
25. Any other co-existing medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent
26. Absence of caregivers in non-autonomous patients
27. Need of anticoagulation with warfarin or another vitamin K antagonist
28. Vaccination with live vaccine within 28 days prior to investigation treatment
29. Have a known hypersensitivity to any of the excipients of Pirtobrutinib or to any intended study medications

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 48 months
  PFS defined as the time between the start of treatment and the first documentation of recurrence, progression or death for any cause

SECONDARY OUTCOMES:
Overall response rate (ORR) | 48 months
  Overall Response Rate (ORR) will be defined as the proportion of patients achieving either a Complete Response (CR) or a Partial Response (PR), according to the Lugano 2014 criteria for response assessment in lymphoma.
Complete response rate (CRR) | 48 months
  Complete response rate (CRR) refers to the proportion of patients whose disease completely disappears following treatment, as determined by clinical, imaging, or pathological assessments. It indicates a full remission of detectable disease.
Overall survival (OS) | 48 months
  Overall survival (OS) is defined as the time between the start of treatment and death from any cause
Event free survival (EFS) | 48 months
  Event free survival (EFS) is defined as the time between the start of treatment and treatment failure including disease progression, or discontinuation of treatment for any reason (e.g., disease progression, toxicity, patient preference, initiation of new treatment without documented progression, or death).
Duration of response (DOR) | 48 months
  Duration of response (DOR) is defined as the time from the first documentation of tumor response to disease progression or death from any cause.
Drop-out rate | 48 months
  Proportion of participants who withdraw from the study for any reason before completing the planned treatment/intervention period.
Rate of treatment discontinuation due to Adverse Event (AE) or treatment intolerance. | 48 months
  Proportion of participants who permanently discontinue the assigned treatment due to adverse events (AEs) or treatment intolerance during the study period.
Frequency and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 48 months
  Frequency and severity of AEs and SAEs classified as per latest version of CTCAE
Health-Related Quality of Life Assessed by the EuroQol 5-Dimension 5-Level (EQ-5D-5L) Questionnaire | 48 months
  The EQ-5D-5L is a standardized instrument for measuring generic health status. It includes five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with five levels. The outcome will be reported as the EQ-5D-5L index score. Higher scores indicate better health status.
Health-Related Quality of Life Assessed by the Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) Questionnaire | 48 months
  The FACT-Lym is a disease-specific instrument assessing quality of life in patients with lymphoma. It includes physical, social/family, emotional, and functional well-being, plus lymphoma-specific concerns. The outcome will be reported as the total FACT-Lym score. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Visco, Prof., Principal Investigator — Verona - AOU Integrata di Verona - U.O. Ematologia; Guido Gini, Dott., Principal Investigator — Ancona - AOU Ospedali Riuniti - Clinica di Ematologia
Locations (20):
- Italy (20):
  - IRCCS Istituto Romagnolo per lo studio dei Tumori "Dino Amadori" - IRST S.R.L. - Ematologia, Meldola, Forlì-Cesena
  - Istituto Clinico Humanitas - U.O. Ematologia, Rozzano, Milano
  - AOU Ospedali Riuniti - Clinica di Ematologia, Ancona
  - Azienda Ospedaliera S.Giuseppe Moscati - S.C. Ematologia e Trapianto emopoietico, Avellino
  - Nuovo Ospedale degli Infermi - SSD Ematologia, Biella
  - Policlinico S.Orsola-Malpighi - Istituto di Ematologia "Seragnoli", Bologna
  - ASST Spedali Civili di Brescia - Ematologia, Brescia
  - Azienda Ospedaliera Universitaria Policlinico - S. Marco - UOC di Ematologia, Catania
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano - Ematologia, Milan
  - A.O. Ospedali Riuniti Villa Sofia-Cervello - Divisione di Ematologia, Palermo
  - Parma - AOU di Parma - UOC Ematologia e CTMO, Parma
  - P.O. Spirito Santo di Pescara - UOC Ematologia Dipartimento Oncologico Ematologico - ASL Pescara, Pescara
  - Azienda USL Piacenza - UOC Ematologia e Centro Trapianti, Piacenza
  - Azienda Unitа Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova - Ematologia, Reggio Emilia
  - AOU Senese - U.O.C. Ematologia, Siena
  - A.O. S. Maria di Terni - S.C. Oncoematologia, Terni
  - Ospedale Ca Foncello - S.C di Ematologia, Treviso
  - Ospedale di Circolo - U.O.C Ematologia, Varese
  - AOU Integrata di Verona - U.O. Ematologia, Verona
  - Vicenza - ULSS 8 Berica - Ospedale S. Bortolo - Ematologia, Vicenza

IPD SHARING:
Plan to Share IPD: Yes
No identifiable data, such as name, address, hospital name, date of birth, or any other identifying data, will be shared and should not be requested. For each data sharing request, it is essential that a proforma (available on request) is completed that describes the general purpose, specific aims, data items requested, analysis plan and acknowledgment of the trial management team. Requests will be reviewed based on scientific merit and ethical principles. Requestors who are granted access to the data will be required to complete a data sharing agreement that will be signed by the requester and FIL. In compliance with the national ethics guideline and applicable legislation, individual deidentified patients' data (including study protocol, statistical analysis plan and data coding) can be shared until 5 years after the publication of the study.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: In compliance with the domestic ethics guideline and applicable legislation, individual deidentified patients' data underlying the results reported in the publication article (including study protocol, statistical analysis plan and data coding) can be shared until 5 years after the publication of the article.
Access Criteria: For each data sharing request, it is essential that a proforma (available on request) is completed that describes the general purpose, specific aims, data items requested, analysis plan and acknowledgment of the trial management team. Requests will be reviewed based on scientific merit and ethical principles. Requestors who are granted access to the data will be required to complete a data sharing agreement that will be signed by the requester and FIL.